CLINICAL TRIAL: NCT01994044
Title: Treating Selected Chronic WAD Patients: Cervical Fusion or Multidimensional Rehabilitation. A Randomized Study
Brief Title: Randomized WAD Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Surgery Clinic, Strängnäs (Other)
Responsible Party: Principal Investigator, Bo Nyström, MD, PhD, Spinal Surgery Clinic, Strängnäs
Purpose: Treatment
Other Study IDs: RKSWAD SpinalSC; SpinalSC (Other: SpinalSC)
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Whiplash Symptoms
Keywords: Whiplash, surgery, multimodal rehabilitation, independent examiners
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multimodal rehabilitation (Active Comparator)
  Interventions: Procedure: Cervical fusion
- Cervical fusion (Active Comparator)
  Interventions: Procedure: Cervical fusion

INTERVENTIONS:
Procedure: Cervical fusion

SUMMARY:
Background: The majority of patients suffering a whiplash injury (WAD) will recover, but some may have symptoms for years despite all kinds of conservative treatment. The Neck Pain Task Force (2008) found no existing evidence for positive effects of fusion operations in such patients. Some of them, however, present with symptoms that might indicate pain from a motion segment, possibly the disc. Our aim was therefore to test this possibility by performing a randomized study comparing cervical fusion and multimodal rehabilitation in chronic WAD patients.

Methods: Patients with a specified symptomatology, all with pronounced symptoms for long periods of time, were recruited and randomized to surgery (25 pat.) or to multimodal rehabilitation (24 pat.). All patients were investigated before start of the study and at follow-up approximately two years after treatment by four independent examiners from disciplines usually involved in treating WAD patients. The patients also gave their own assessments of the treatment results. Seven patients in each group did not undergo the allocated treatment for various reasons.

DETAILED DESCRIPTION:
Outcomes:

representing different disciplines: neurology, orthopedics, physical medicine and psychology. Each patient´s perceived change in outcome was also assessed. Assessment was made before treatment and at follow-up two years afterwards.

In addition to the assessments of outcome made by the examiners, the patients completed the SF-36, EQ-5D and BIS (Balanced Inventory for Spinal Disorders) questionnaires before treatment and at follow-up. The results of these assessments will be given in a forthcoming paper.

6b. No changes in trial outcomes were made during the study.

ELIGIBILITY:
Inclusion Criteria:

* The patients were to have been involved in a traffic accident as the origin of their pain and to have had pronounced symptoms lasting for at least one year.
* They should be in the age group 18 to 60 years,
* have been actively working up until the accident,
* should not have had previous neck pain.
* All patients should have had a plain X-ray and an MRI showing no specific changes.
* The patients should present with pronounced neck pain with the origin in the midline.
* The character of the pain should be dull, aching, and, with sudden movements, stabbing in the same area.
* Palpation and pressure in that area should provoke deep pain..

Exclusion Criteria:

- Previous pain in the neck, previous surgery

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 1999-07; Primary Completion 2005-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Complaints of WAD | Independent examiners
SF-36 questionnaire | Follow-up at 2 years

SECONDARY OUTCOMES:
Complaints of WAD | SF-36
Range of neck movement | Follow-up at 2 years

OTHER OUTCOMES:
Complaints of WAD | BIS (Balanced Inventory for Spinal Disorders)
Quality of Life (Balanced Inventory for Spinal Disorders, questionnaire) | Follow-up at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bo Nyström, MD, PhD, Principal Investigator — Clinic of Spinal Surgery
Locations (1):
- Clinic of Spinal Surgery, Strängnäs, Sweden

REFERENCES:
- [Background] Carragee EJ, Hurwitz EL, Cheng I, Carroll LJ, Nordin M, Guzman J, Peloso P, Holm LW, Cote P, Hogg-Johnson S, van der Velde G, Cassidy JD, Haldeman S; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Treatment of neck pain: injections and surgical interventions: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S153-69. doi: 10.1097/BRS.0b013e31816445ea. PMID 18204388
- See also: Related Info — http://www.ryggkirurgiska.se